CLINICAL TRIAL: NCT01724021
Title: A Randomized, Open-label, Mutli-centre Study to Evaluate Patient Preference With Subcutaneous Administration of Rituximab Versus Intravenous Rituximab in Previously Untreated Patients With CD20+ Diffuse Large B-cell Lymphoma or CD20+ Follicular Non-Hodgkin's Lymphoma Grades 1, 2, OR 3A
Brief Title: A Study of Participant Preference With Subcutaneous Versus Intravenous MabThera/Rituxan in Participants With CD20+ Diffuse Large B-Cell Lymphoma or CD20+ Follicular Non-Hodgkin's Lymphoma Grades 1, 2 or 3a
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO28457; 2012-003230-17 (EudraCT Number)
Record Dates: First submitted 2012-11-05; First posted 2012-11-09 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Diffuse Large B-Cell Lymphoma, Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Prednisolone; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Participants in Arm A received one cycle of rituximab 375 mg/m^2 intravenously (IV), then three cycles of rituximab 1400mg subcutaneously (SC), followed by four cycles of rituximab 375 mg/m^2 IV in combination with a standard chemotherapy of cyclophosphamide, hydroxydaunorubicin, Oncovin, prednisone/prednisolone (CHOP), cyclophosphamide, vincristine, prednisone/prednisolone (CVP), or bendamustine. Rituximab was administered on Day 1 of each treatment cycle followed by administration of the preselected chemotherapy. Cycles were repeated every 14, 21, or 28 days, depending on the combination chemotherapy regimen selected by the investigator.
  Interventions: Drug: Cyclophosphamide, Hydroxydaunorubicin, Oncovin, Prednisone/Prednisolone (CHOP); Drug: Cyclophosphamide, Vincristine, Prednisone/Prednisolone (CVP); Drug: Bendamustine; Drug: Rituximab
- Arm B (Experimental): Participants in Arm B received four cycles of rituximab 375 mg/m^2 IV followed by four cycles of rituximab 1400mg SC in combination with a standard chemotherapy of CHOP, CVP, or bendamustine. Rituximab was administered on Day 1 of each treatment cycle followed by administration of the preselected chemotherapy. Cycles were repeated every 14, 21, or 28 days, depending on the combination chemotherapy regimen selected by the investigator.
  Interventions: Drug: Cyclophosphamide, Hydroxydaunorubicin, Oncovin, Prednisone/Prednisolone (CHOP); Drug: Cyclophosphamide, Vincristine, Prednisone/Prednisolone (CVP); Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Cyclophosphamide, Hydroxydaunorubicin, Oncovin, Prednisone/Prednisolone (CHOP) — Standard chemotherapy
Drug: Cyclophosphamide, Vincristine, Prednisone/Prednisolone (CVP) — Standard chemotherapy
Drug: Bendamustine — Standard chemotherapy
  Other Names: Treanda
Drug: Rituximab — 1400 mg subcutaneously (SC), Day 1 Cycles 2-4
  Other Names: Rituxan; MabThera
  Arms: Arm A
Drug: Rituximab — 375 mg/m2 IV, Day 1 Cycles 1-4
  Other Names: Rituxan; MabThera
  Arms: Arm B
Drug: Rituximab — 375 mg/m2 intravenously (IV), Day 1 Cycles 1 and 4-8
  Other Names: Rituxan; MabThera
  Arms: Arm A
Drug: Rituximab — 1400 mg SC, Day 1 Cycles 5-8
  Other Names: Rituxan; MabThera
  Arms: Arm B

SUMMARY:
This multi-center, open-label, randomized study will evaluate the participant preference with subcutaneous versus intravenous administration of MabThera/Rituxan (rituximab) in participants with CD20+ diffuse large B-cell lymphoma or CD20+ follicular non-Hodgkin's lymphoma. In Arm A, participants will receive MabThera/Rituxan 375 mg/m2 intravenously (IV) on Day 1 of Cycle 1 and MabThera/Rituxan 1400 mg subcutaneously (SC) on Day 1 of Cycles 2-4, followed by MabThera/Rituxan IV in Cycles 5-8. Participants in Arm B will receive MabThera/Rituxan IV in Cycles 1-4 and SC in Cycles 5-8. All participants will receive 6-8 cycles of standard chemotherapy (according to local country practice) with 8 cycles of MabThera/Rituxan. Anticipated time on study treatment is up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants , >/= 18 and </= 80 years of age
* Histologically confirmed, previously untreated CD20+ diffuse large B-cell lymphoma (DLBCL) or CD20+ follicular non-Hodgkin's lymphoma (NHL) Grade 1, 2, or 3a, according to World Health Organization (WHO) classification
* An International Prognostic Index (IPI) score of 1-4 or IPI score of 0 with bulky disease, defined as one lesion >/= 7.5 cm, or Follicular Lymphoma International Prognostic Index (FLIPI; low, intermediate or high risk)
* At least one bi-dimensionally measurable lesion defined as >/=1.5 cm in its largest dimension on CT scan
* Eastern Cooperative Oncology Group (ECOG) performance status </= 3

Exclusion Criteria:

* Transformed lymphoma or follicular lymphoma IIIB
* Primary central nervous system (CNS) lymphoma, histologic evidence of transformation to Burkitt lymphoma, primary mediastinal DLBCL, primary effusion lymphoma, primary cutaneous DLBCL, or primary DLBCL of the testis
* History of other malignancy that could affect compliance with the protocol or interpretation of the results; this includes a malignancy that has been treated but not with curative intent, unless the malignancy has been in remission for >/= 5 years prior to enrolment; participants with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix are eligible
* Prior therapy for DLBCL or NHL, with the exception of nodal biopsy or local irradiation
* Prior treatment with cytotoxic drugs (with the exclusion of intrathecal methotrexate for CNS prophylaxis in DLBCL) or rituximab for another condition, or prior use of an anti-CD20 drug
* Prior use of monoclonal antibody within 3 months prior to randomization
* Chemotherapy or other investigational therapy within 28 days prior to randomization
* Ongoing corticosteroid use > 30 mg/day prednisolone or equivalent
* Inadequate renal. hematologic or hepatic function
* Active and/or severe infection or any major episode of infection within 4 weeks prior to randomization
* Active hepatitis B virus or active hepatitis C virus infection
* History of human immunodeficiency (HIV) seropositive status
* A positive pregnancy test in women of childbearing potential
* Life expectancy of less than 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 743 (Actual)
Dates: Start 2012-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (214):
- Argentina (3):
  - Buenos Aires
  - Corrientes
  - Santa Fé
- Australia (13):
  - Canberra, Australian Capital Territory
  - Camperdown, New South Wales
  - Liverpool, New South Wales
  - Randwick, New South Wales
  - Brisbane, Queensland
  - Adelaide, South Australia
  - Hobart, Tasmania
  - Geelong, Victoria
  - Malvern, Victoria
  - Melbourne, Victoria
  - Wodonga, Victoria
  - Nedlands, Western Australia
  - Perth, Western Australia
- Austria (5):
  - Krems
  - Linz
  - Salzburg
  - Steyr
  - Vienna
- Brazil (11):
  - Belo Horizonte, Minas Gerais
  - Juiz de Fora, Minas Gerais
  - Varginha, Minas Gerais
  - Curitiba, Paraná
  - Londrina, Paraná
  - Recife, Pernambuco
  - Caxias do Sul, Rio Grande do Sul
  - Novo Hamburgo, Rio Grande do Sul
  - Santa Maria, Rio Grande do Sul
  - Santo André, São Paulo
  - São José do Rio Preto, São Paulo
- Canada (5):
  - Burnaby, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Hamilton, Ontario
  - Montreal, Quebec
- Chile (2):
  - Santiago
  - Viña del Mar
- Montería, Colombia
- Osijek, Croatia
- Denmark (2):
  - Aalborg
  - Holstebro
- Santiago de los Caballeros, Dominican Republic
- Egypt (2):
  - Alexandria
  - Cairo
- San Salvador, El Salvador
- Germany (83):
  - Aschaffenburg
  - Augsburg
  - Bamberg
  - Bayreuth
  - Berlin
  - Bielefeld
  - Bochum
  - Bonn
  - Bottrop
  - Brandenburg
  - Bremen
  - Bremerhaven
  - Coesfeld
  - Cologne
  - Darmstadt
  - Dresden
  - Düsseldorf
  - Eisenach
  - Essen
  - Frankfurt
  - Frankfurt (Oder)
  - Freiburg im Breisgau
  - Fürth
  - Georgsmarienhütte
  - Giessen
  - Goslar
  - Gütersloh
  - Halle
  - Hamburg
  - Hamm
  - Hanau
  - Hanover
  - Herford
  - Jena
  - Kaiserslautern
  - Kassel
  - Leer
  - Leipzig
  - Limburg
  - Lübeck
  - Magdeburg
  - Mainz
  - Mannheim
  - Marburg
  - Mayen
  - Moers
  - Mönchengladbach
  - Mutlangen
  - Mülheim
  - München
  - Münster
  - Neunkirchen/Saar
  - Nuremberg
  - Oldenburg
  - Osnabrück
  - Paderborn
  - Pforzheim
  - Pinneberg
  - Pirna
  - Porta Westfalica
  - Pößneck
  - Ravensburg
  - Recklinghausen
  - Regensburg
  - Rostock
  - Rötha
  - Schwäbisch Hall
  - Schweinfurt
  - Siegburg
  - Stade
  - Stendal
  - Stuttgart
  - Traunstein
  - Trier
  - Velbert
  - Villingen-Schwenningen
  - Weilheim
  - Wiesbaden
  - Wilhelmshaven
  - Witten
  - Würselen
  - Zittau
  - Zwickau
- Guatemala City, Guatemala
- Hong Kong, Hong Kong
- Hungary (7):
  - Budapest
  - Győr
  - Gyula
  - Kaposvár
  - Nyíregyháza
  - Szeged
  - Szolnok
- Indonesia (4):
  - Bandung
  - Jakarta
  - Surabaya
  - Yogyakarta
- Italy (12):
  - Brindisi, Apulia
  - Lecce, Apulia
  - Catanzaro, Calabria
  - Ferrara, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Piacenza, Emilia-Romagna
  - Rome, Lazio
  - Candiolo, Piedmont
  - Cuneo, Piedmont
  - Palermo, Sicily
  - Lido di Camaiore, Tuscany
  - Livorno, Tuscany
- Malaysia (4):
  - Ampang
  - Kuala Lumpur
  - Kuching
  - Sabak Bernam
- Netherlands (13):
  - Amstelveen
  - Amsterdam
  - Apeldoorn
  - Beverwijk
  - Capelle aan den IJssel
  - Delftzijl
  - Eindhoven
  - Goes
  - Leidschendam
  - Rotterdam
  - The Hague
  - Tilburg
  - Utrecht
- Auckland, New Zealand
- Panama City, Panama
- Peru (3):
  - Arequipa
  - Cusco
  - La Victoria, Lima
- Philippines (3):
  - Cebu City
  - Manila
  - Quezon City
- Portugal (5):
  - Lisbon
  - Matosinhos Municipality
  - Ponta Delgada
  - Setúbal
  - Viseu
- Romania (8):
  - Baia Mare
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Iași
  - Sibiu
  - Timișoara
- South Korea (3):
  - Busan
  - Daegu
  - Seoul
- Sweden (6):
  - Falun
  - Gothenburg
  - Jönköping
  - Karlstad
  - Sundsvall
  - Västerås
- Taiwan (3):
  - Kaohsung
  - Taichung
  - Taipei
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
- Turkey (Türkiye) (4):
  - Ankara
  - Denizli
  - Erzurum
  - Malatya
- Vietnam (2):
  - Hà Nội
  - Hochiminh City

REFERENCES:
- [Derived] Rummel M, Kim TM, Aversa F, Brugger W, Capochiani E, Plenteda C, Re F, Trask P, Osborne S, Smith R, Grigg A. Preference for subcutaneous or intravenous administration of rituximab among patients with untreated CD20+ diffuse large B-cell lymphoma or follicular lymphoma: results from a prospective, randomized, open-label, crossover study (PrefMab). Ann Oncol. 2017 Apr 1;28(4):836-842. doi: 10.1093/annonc/mdw685. PMID 28031173
- [Derived] Theodore-Oklota C, Humphrey L, Wiesner C, Schnetzler G, Hudgens S, Campbell A. Validation of a treatment satisfaction questionnaire in non-Hodgkin lymphoma: assessing the change from intravenous to subcutaneous administration of rituximab. Patient Prefer Adherence. 2016 Sep 13;10:1767-1776. doi: 10.2147/PPA.S108489. eCollection 2016. PMID 27695295

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 743 participants were enrolled across all the sites and were included in the intent to treat (ITT) population. Three participants were enrolled but died prior to receiving study medication and were not included in the safety population. The Participant Flow represents the safety population.
Groups:
- Arm A: Participants in Arm A received one cycle of rituximab 375 milligram per metre square (mg/m^2) intravenously (IV), then three cycles of rituximab 1400mg subcutaneously (SC), followed by four cycles of rituximab 375 mg/m^2 IV in combination with a standard chemotherapy of cyclophosphamide, hydroxydaunorubicin, Oncovin, prednisone/prednisolone (CHOP), cyclophosphamide, vincristine, prednisone/prednisolone (CVP), or bendamustine. Rituximab was administered on Day 1 of each treatment cycle followed by administration of the preselected chemotherapy. Cycles were repeated every 14, 21, or 28 days, depending on the combination chemotherapy regimen selected by the investigator.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 371 | 369
Completed | 244 | 236
Not Completed | 127 | 133
Not completed — Adverse Event | 11 | 6
Not completed — Death | 46 | 58
Not completed — Participant request/ Withdrew consent | 18 | 14
Not completed — Lost to Follow-up | 15 | 15
Not completed — Reason Not Specified | 36 | 39
Not completed — Missing | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 371 | 369 | 740
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (13.18) | 59.4 (12.64) | 58.8 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 180 | 367
  Male | 184 | 189 | 373

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Indicating a Preference for Rituximab Subcutaneous (SC) Over Rituximab Intravenously (IV) at Cycle 6
Description: Participants who preferred rituximab SC over rituximab IV, along with the corresponding 95% confidence interval (CI), were estimated using the patient preference questionnaire (PPQ) after completing cycle 6.
Time Frame: Cycle 6 (Up to 24 weeks)
Population: ITT population included all participants who were randomized in the study. Number of participants analyzed specifies number of participants who were evaluable for the outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 372 | 371
percentage of participants | 79.1 [74.2 to 83.5] | 80.6 [75.7 to 84.8]

2. Primary Outcome: Percentage of Participants Indicating a Preference for Rituximab Subcutaneous (SC) Over Rituximab Intravenously (IV) at Cycle 8
Description: Participants who preferred rituximab SC over rituximab IV, along with the corresponding 95% confidence interval (CI), were estimated using the patient preference questionnaire (PPQ) after completing Cycle 8.
Time Frame: Cycle 8 (Up to 32 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 372 | 371
percentage of participants | 77.1 [71.9 to 81.8] | 84.2 [79.6 to 88.2]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Randomization of first participant to clinical cutoff date (Up to 4 years)
Population: The safety population included all participants who received at least one dose of rituximab. Number of participants analyzed specifies number of participants who were evaluable for the outcome measure.
Measure: Number; unit: participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 371 | 369
participants | 352 | 347

4. Secondary Outcome: Time Required for Rituximab Administration (Subcutaneous [SC] or Intravenous [IV])
Description: Administration time was defined as the time from start to end of the SC injection or from start to end of the IV infusion
Time Frame: Cycle 1-4, Cycle 5-8 for both SC and IV (Up to 32 weeks)
Population: ITT population included all participants who were randomized in the study.
Measure: Median (Full Range); unit: minutes
Groups:
- Rituximab Intravenous (IV): Rituximab was administered at a dose of 375 mg/m2 body surface area (BSA) as a single IV infusion, followed by administration of chemotherapy. At Cycle 1, Day 1, the first rituximab dose for both Arms A and B was always administered as a slow IV infusion, according to local standard practice. Faster infusion rates were permitted after Cycle 1, according to local practice. Cycles were repeated every 14, 21, or 28 days, depending on the combination chemotherapy regimen selected by the investigator.
- Rituximab Subcutaneous (SC): Each treatment cycle consisted of a single SC injection of rituximab administered at a fixed dose of 1400 mg. Rituximab was administered on Day 1 of each treatment cycle followed by administration of the preselected chemotherapy. Cycles were repeated every 14, 21, or 28 days, depending on the combination chemotherapy regimen selected by the investigator.
Arm/Group | Rituximab Intravenous (IV) | Rituximab Subcutaneous (SC)
Number analyzed (Participants) | 740 | 687
minutes | 840 [0 to 3967.0] | 22 [0 to 1242.0]

5. Secondary Outcome: Cancer Therapy Satisfaction Questionnaire (CTSQ) Score
Description: CTSQ is a validated 16-item questionnaire that measures three domains related to participants' satisfaction with cancer therapy. These include expectations of therapy, feelings about side effects, and satisfaction with therapy. Each domain is scored on a scale of 0 to 100, with higher scores indicative of more positive feelings toward therapy. The score for each domain was averaged among all participants.
Time Frame: During Cycle 4, 8 of treatment (Up to 32 weeks)
Population: ITT population included all participants who were randomized in the study. Here, "Number Analyzed" represents the number of participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab Intravenous (IV) | Rituximab Subcutaneous (SC)
Number analyzed (Participants) | 740 | 687
units on a scale
  Expectations of therapy domain: number analyzed (Participants) | 631 | 627
  Expectations of therapy domain | 80.88 (18.315) | 82.07 (17.817)
  Feelings about side effects domain: number analyzed (Participants) | 630 | 624
  Feelings about side effects domain | 60.63 (22.316) | 61.64 (22.324)
  Satisfaction with therapy domain: number analyzed (Participants) | 619 | 623
  Satisfaction with therapy domain | 84.59 (12.218) | 85.42 (11.259)

6. Secondary Outcome: Rituximab Administration Satisfaction Questionnaire (RASQ) Score
Description: The RASQ is a 20-item questionnaire that measures five domains related to the impact of treatment administration. These include physical impact, psychological impact, impact on activities of daily living (ADLs), convenience, and satisfaction. Each domain is scored on a scale of 0 to 100, with higher scores indicative of more positive feelings toward therapy. The score for each domain was averaged among all participants.
Time Frame: During Cycle 4, 8 of treatment (Up to 32 weeks)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rituximab Intravenous (IV) | Rituximab Subcutaneous (SC)
Number analyzed (Participants) | 740 | 687
units on a scale
  Physical impact domain: number analyzed (Participants) | 622 | 618
  Physical impact domain | 82.14 (15.629) | 82.08 (15.882)
  Psychological Impact domain: number analyzed (Participants) | 614 | 612
  Psychological Impact domain | 77.73 (16.377) | 84.00 (14.358)
  Impact on activitiesf daily living: number analyzed (Participants) | 604 | 600
  Impact on activitiesf daily living | 59.49 (22.233) | 81.86 (15.844)
  Convenience domain: number analyzed (Participants) | 620 | 599
  Convenience domain | 59.05 (20.757) | 81.05 (13.088)
  Satisfaction domain: number analyzed (Participants) | 617 | 624
  Satisfaction domain | 74.88 (19.349) | 87.26 (14.972)

7. Secondary Outcome: Complete Response (CR) Rate
Description: CR rate was assessed according to the International Working Group (IWG) Response Criteria (CHESON ET AL. 1999) and included CR and CR unconfirmed (CRu). CR was defined as complete disappearance of all clinical and radiographic evidence of disease and disease-related symptoms, regression of lymph nodes to normal size, absence of splenomegaly, and absence of bone marrow involvement. CRu was defined as disappearance of clinical and radiographic evidence of disease and absence of splenomegaly, with regression of lymph nodes by > 75 % but still >1.5 cm in size, and indeterminate bone marrow assessment. Tumor assessments were based on computed tomography (CT) scans with contrast of the neck, chest, and abdomen (if detectable by these techniques) or other diagnostic means, if applicable. Other methods (e.g., MRI) were acceptable for participants in whom contrast CT scans were contraindicated. Due to the limited availability of FDG-PET scanners, an FDG-PET scan was not mandated in the study.
Time Frame: 28 days (± 3 days) after Day 1 of the last dose of induction treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 307 | 315
percentage of participants | 49.2 [43.5 to 54.9] | 52.7 [47.0 to 58.3]

8. Secondary Outcome: Event-free Survival (EFS)
Description: EFS was defined as the time from randomization to first occurrence of progression or relapse according to IWG response criteria. IWG criteria is defined using the following response categories: CR: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy; partial response (PR): At least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses; stable disease (SD): participants fails to attain the criteria needed for a CR or PR, but does not fulfill those for progressive disease (PD); PD: Lymph nodes considered abnormal if the long axis is more than 1.5 centimeter (cm) regardless of the short axis. Lymph node has a long axis of 1.1 to 1.5 cm, it is considered abnormal if its short axis is more than 1.0. Lymph nodes less than or equal to (<=) 1.0 × <= 1.0 cm would not be considered as abnormal for PD.
Time Frame: From the time of randomization until disease progression or 24 months post treatment follow up or which ever occur first (Up to 4 years)
Population: ITT population included all participants who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 372 | 371
months | NA [NA to NA] — Median (and it's CI) was not reached for this Outcome Measure. | NA [NA to NA] — Median (and it's CI) was not reached for this Outcome Measure.

9. Secondary Outcome: Disease-free Survival (DFS)
Description: DFS was defined as the period from the data of the initial CR/CRu until the date of relapse or death from any cause, whichever occurred first.
Time Frame: as for outcome 8
Population: ITT population included all participants who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 372 | 371
months | NA [NA to NA] — Median (and it's CI) was not reached for this Outcome Measure. | NA [NA to NA] — Median (and it's CI) was not reached for this Outcome Measure.

10. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to the first occurrence of progression or relapse, according to the IWG response criteria. IWG criteria is defined criteria using the following response categories: CR: Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy; PR: At least a 50% decrease in SPD of up to six of the largest dominant nodes or nodal masses; SD: participants fails to attain the criteria needed for a CR or PR, but does not fulfill those for PD; PD: Lymph nodes considered abnormal if the long axis is more than 1.5 cm regardless of the short axis. Lymph node has a long axis of 1.1 to 1.5 cm, it is considered abnormal if its short axis is more than 1.0. Lymph nodes <= 1.0 × <= 1.0 cm would not be considered as abnormal for PD.
Time Frame: as for outcome 8
Population: ITT population included all participants who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 372 | 371
months | NA [NA to NA] — Median (and it's CI) was not reached for this Outcome Measure. | NA [NA to NA] — Median (and it's CI) was not reached for this Outcome Measure.

11. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: as for outcome 8
Population: ITT population included all participants who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 372 | 371
months | NA [NA to NA] — Median (and it's CI) was not reached for this Outcome Measure. | NA [NA to NA] — Median (and it's CI) was not reached for this Outcome Measure.

12. Secondary Outcome: Percentage of Participants With Anti-Rituximab Antibodies Over Time
Time Frame: Pre-dose Cycle 1 to 8, interim staging, final staging, 6, 12 months follow-up, end of study (Up to 4 years)
Population: The safety population included all participants who received at least one dose of rituximab. Here, "Number Analyzed" represents the number of participants who were evaluable at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 371 | 369
percentage of participants
  Cycle 1: number analyzed (Participants) | 342 | 335
  Cycle 1 | 2.0 | 3.0
  Cycle 2: number analyzed (Participants) | 333 | 325
  Cycle 2 | 2.1 | 2.2
  Cycle 3: number analyzed (Participants) | 328 | 322
  Cycle 3 | 0.3 | 0.9
  Cycle 4: number analyzed (Participants) | 323 | 323
  Cycle 4 | 0 | 0.3
  Interim staging: number analyzed (Participants) | 283 | 281
  Interim staging | 0 | 0
  Cycle 5: number analyzed (Participants) | 237 | 253
  Cycle 5 | 0 | 0
  Cycle 6: number analyzed (Participants) | 300 | 289
  Cycle 6 | 0 | 0
  Cycle 7: number analyzed (Participants) | 288 | 290
  Cycle 7 | 0 | 0
  Cycle 8: number analyzed (Participants) | 281 | 283
  Cycle 8 | 0 | 0
  Final staging: number analyzed (Participants) | 261 | 260
  Final staging | 0 | 0
  Follow-up, 6 months: number analyzed (Participants) | 166 | 183
  Follow-up, 6 months | 1.8 | 0
  Follow-up, 12 months: number analyzed (Participants) | 141 | 161
  Follow-up, 12 months | 2.1 | 0.6
  End of study/early treatment termination: number analyzed (Participants) | 174 | 171
  End of study/early treatment termination | 0.6 | 0.6

13. Secondary Outcome: Percentage of Participants With Anti-Recombinant Human Hyaluronidase (rHuPH20) Antibodies Over Time
Time Frame: Pre-dose Cycle 1 to 8, interim staging, final staging, 6, 12 months follow-up, end of study (Up to 4 years)
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 371 | 369
percentage of participants
  Cycle 1: number analyzed (Participants) | 35 | 32
  Cycle 1 | 11.4 | 15.6
  Cycle 2: number analyzed (Participants) | 342 | 33
  Cycle 2 | 7.0 | 18.2
  Cycle 3: number analyzed (Participants) | 339 | 34
  Cycle 3 | 7.1 | 23.5
  Cycle 4: number analyzed (Participants) | 327 | 34
  Cycle 4 | 7.0 | 14.7
  Interim staging: number analyzed (Participants) | 279 | 269
  Interim staging | 9.0 | 9.7
  Cycle 5: number analyzed (Participants) | 24 | 266
  Cycle 5 | 12.5 | 10.2
  Cycle 6: number analyzed (Participants) | 25 | 303
  Cycle 6 | 16.0 | 11.6
  Cycle 7: number analyzed (Participants) | 21 | 303
  Cycle 7 | 23.8 | 10.9
  Cycle 8: number analyzed (Participants) | 15 | 291
  Cycle 8 | 13.3 | 11.0
  Final staging: number analyzed (Participants) | 240 | 261
  Final staging | 10.0 | 12.6
  Follow-up, 6 months: number analyzed (Participants) | 155 | 172
  Follow-up, 6 months | 6.5 | 13.4
  Follow-up, 12 months: number analyzed (Participants) | 142 | 161
  Follow-up, 12 months | 7.7 | 8.7
  End of study/early treatment termination: number analyzed (Participants) | 171 | 175
  End of study/early treatment termination | 3.5 | 6.3

14. Secondary Outcome: Summary of Observed Serum Rituximab Concentration
Time Frame: Pre-dose Cycle 1 to 8, interim staging, final staging, 6, 12 months follow-up, end of study (Up to 4 years)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: microgram per milliter
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 371 | 369
microgram per milliter
  Cycle 1: number analyzed (Participants) | 285 | 281
  Cycle 1 | 3355.9 (21600.95) | 970.1 (9415.93)
  Cycle 2: number analyzed (Participants) | 284 | 280
  Cycle 2 | 25053.1 (19590.17) | 24541.1 (18141.76)
  Cycle 3: number analyzed (Participants) | 281 | 281
  Cycle 3 | 62977.0 (30037.98) | 46093.9 (31214.30)
  Cycle 4: number analyzed (Participants) | 282 | 285
  Cycle 4 | 87956.6 (40441.84) | 59485.5 (29183.17)
  Interim staging: number analyzed (Participants) | 256 | 251
  Interim staging | 117273.6 (52227.06) | 77665.3 (29161.77)
  Cycle 5: number analyzed (Participants) | 212 | 226
  Cycle 5 | 108030.9 (54335.08) | 70387.3 (30256.48)
  Cycle 6: number analyzed (Participants) | 282 | 266
  Cycle 6 | 100927.7 (49287.42) | 98679.7 (40001.55)
  Cycle 7: number analyzed (Participants) | 272 | 268
  Cycle 7 | 95614.0 (45499.56) | 117172.0 (44501.74)
  Cycle 8: number analyzed (Participants) | 267 | 266
  Cycle 8 | 104873.0 (50346.69) | 137048.1 (53669.39)
  Final staging: number analyzed (Participants) | 253 | 252
  Final staging | 86806.6 (43005.90) | 120995.7 (58731.10)
  Follow-up, 6 months: number analyzed (Participants) | 164 | 183
  Follow-up, 6 months | 7802.9 (15672.57) | 8042.9 (12247.05)
  Follow-up, 12 months: number analyzed (Participants) | 139 | 163
  Follow-up, 12 months | 2380.1 (8494.06) | 1685.3 (6669.84)
  End of study/early treatment termination: number analyzed (Participants) | 173 | 168
  End of study/early treatment termination | 9302.0 (27234.88) | 9553.9 (30723.30)

ADVERSE EVENTS:
Time Frame: Randomization of first participant to clinical cutoff date (Up to 4 years)
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 126/371 | 116/369
Other Adverse Events (participants affected / at risk) | 318/371 | 317/369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=371) | Arm B (N=369)
Febrile Neutropenia (Blood and lymphatic system disorders) | 31 | 30
Neutropenia (Blood and lymphatic system disorders) | 16 | 13
Anaemia (Blood and lymphatic system disorders) | 3 | 5
Leukopenia (Blood and lymphatic system disorders) | 5 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 2
Pneumonia (Infections and infestations) | 12 | 9
Sepsis (Infections and infestations) | 3 | 5
Lung Infection (Infections and infestations) | 3 | 3
Herpes Zoster (Infections and infestations) | 1 | 3
Urinary Tract Infection (Infections and infestations) | 3 | 3
Septic Shock (Infections and infestations) | 2 | 2
Atypical pneumonia (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 1 | 3
Infection (Infections and infestations) | 3 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 2 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 2 | 0
Pneumonia viral (Infections and infestations) | 1 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 2
Soft tissue infection (Infections and infestations) | 0 | 2
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchopulmonary Aspergillosis (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis Bacterial (Infections and infestations) | 0 | 1
Injection site abscess (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lymph node abscess (Infections and infestations) | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 1
Oral fungal infection (Infections and infestations) | 1 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1
Peritonsillitis (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0
Pyoderma (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 11 | 10
White blood cell count decreased (Investigations) | 3 | 3
Alanine aminotransferase increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Pyrexia (General disorders) | 10 | 3
Asthenia (General disorders) | 4 | 1
General physical health deterioration (General disorders) | 3 | 0
Chest pain (General disorders) | 1 | 0
Injection site warmth (General disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Vith nerve paralysis (Nervous system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypernataemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 1 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 3
Circulatory collapse (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 2
Anaphylactic reaction (Immune system disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Diabetes insipidus (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Adverse drug reaction (General disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Genital infection bacterial (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Systemic infection (Infections and infestations) | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=371) | Arm B (N=369)
Nausea (Gastrointestinal disorders) | 83 | 102
Constipation (Gastrointestinal disorders) | 59 | 60
Vomiting (Gastrointestinal disorders) | 44 | 57
Diarrhoea (Gastrointestinal disorders) | 45 | 50
Stomatitis (Gastrointestinal disorders) | 23 | 23
Abdominal pain (Gastrointestinal disorders) | 23 | 19
Abdominal pain upper (Gastrointestinal disorders) | 17 | 22
Neutropenia (Blood and lymphatic system disorders) | 51 | 70
Anaemia (Blood and lymphatic system disorders) | 79 | 68
Leukopenia (Blood and lymphatic system disorders) | 38 | 32
Fatigue (General disorders) | 69 | 91
Pyrexia (General disorders) | 55 | 48
Mucosal inflammation (General disorders) | 25 | 26
Chills (General disorders) | 29 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 60 | 56
Pruritus (Skin and subcutaneous tissue disorders) | 29 | 17
Rash (Skin and subcutaneous tissue disorders) | 19 | 21
Neuropathy peripheral (Nervous system disorders) | 37 | 47
Headache (Nervous system disorders) | 27 | 29
Paraesthesia (Nervous system disorders) | 18 | 36
Cough (Respiratory, thoracic and mediastinal disorders) | 45 | 38
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 21
Nasopharyngitis (Infections and infestations) | 20 | 19
Upper respiratory tract infection (Infections and infestations) | 22 | 20
Neutrophil count decreased (Investigations) | 63 | 69
White blood cell count decreased (Investigations) | 37 | 33
Decreased appetite (Metabolism and nutrition disorders) | 34 | 32
Insomnia (Psychiatric disorders) | 25 | 31
Oedema peripheral (General disorders) | 17 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.